CLINICAL TRIAL: NCT02502487
Title: Dorsal Penile Nerve Block for Rigid Cystoscopy in Men: a Single-center, Randomized, Double-blind and Placebo-controlled Study
Brief Title: Dorsal Penile Nerve Block for Rigid Cystoscopy in Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Yan Qiu, Attending Physician, West China Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: WestChinaHAesthesia-1
Record Dates: First submitted 2015-07-06; First posted 2015-07-20 (Estimated); Results first posted 2016-07-11 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Pain
Keywords: Analgesia; Cystoscopy; Dorsal nerve of penis; Nerve block; Ropivacaine
MeSH Terms: conditions — Pain; Agnosia | interventions — Ropivacaine; Tetracaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tetracaine gel group (Placebo Comparator): Dorsal penile nerve block with saline and tetracaine gel into urethra before rigid cystoscopy
  Interventions: Drug: Tetracaine
- Dorsal penile nerve block group (Experimental): Dorsal penile nerve block with ropivacaine and plain lubricating gel into urethra before rigid cystoscopy
  Interventions: Procedure: Dorsal Penile Nerve Block; Drug: Ropivacaine
- Combination group (Experimental): Dorsal penile nerve block with ropivacaine and tetracaine gel into urethra before rigid cystoscopy
  Interventions: Procedure: Dorsal Penile Nerve Block; Drug: Ropivacaine; Drug: Tetracaine

INTERVENTIONS:
Procedure: Dorsal Penile Nerve Block — Dorsal penile nerve block with 0.33% ropivacaine using 22-G needle in the sub-pubic space at the base of the penis
  Arms: Combination group; Dorsal penile nerve block group
Drug: Ropivacaine — 0.33% Ropivacaine administered around dorsal penile nerve using 22-G needle in the sub-pubic space at the base of the penis
  Arms: Combination group; Dorsal penile nerve block group
Drug: Tetracaine — 1% Tetracaine gel instilled into urethra
  Arms: Combination group; Tetracaine gel group

SUMMARY:
This study will determine the effectiveness and safety of dorsal penile nerve block (DPNB) in men undergoing rigid cystoscopy.

DETAILED DESCRIPTION:
Pain is common in men undergoing rigid cystoscopy. Even with application of a lubricant containing 2% lidocaine, about 76% men suffer from mild to severe pain when undergoing rigid cystoscopy, and approximately 27% men could still feel mild to moderate pain 7 days after the procedure. The most painful part of the procedure for men is when the cystoscope passes through the membranous urethra. Song et al did autopsy on males found dorsal nerve of the penis (DNP), the terminal branch of the pudendal nerve, innervates the membranous urethra in 53.3% specimens. In addition, urethral mucosa has branches of DNP innervated. Dorsal penile nerve block (DPNB) is usually used for circumcision in children and it has been shown to provide effective analgesia for penile surgeries. According to the evidence that some DNP branches innervate membranous urethra and urethra mucosa and most pain originates from cystoscope passing through membranous urethra, we speculated that DPNB could overall reduce pain level in men during rigid cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) Physical Status I-II
* Without history of urethral or prostatic surgery
* Without respiration or circulation disorders
* Without chronic pain

Exclusion Criteria:

* Allergy to local anesthetics
* Coagulation disorder or usage of antiplatelet drugs
* Infection at the site of puncture point
* Severe urethral stenosis

Ages: 20 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2015-06; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guizhi Du, Doctor, Principal Investigator — West China Hospital of Sichuan University, Department of Anesthesiology
Locations (1):
- West China Hospital of Sichuan University, Department of Anesthesiology, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Babjuk M, Burger M, Zigeuner R, Shariat SF, van Rhijn BW, Comperat E, Sylvester RJ, Kaasinen E, Bohle A, Palou Redorta J, Roupret M; European Association of Urology. EAU guidelines on non-muscle-invasive urothelial carcinoma of the bladder: update 2013. Eur Urol. 2013 Oct;64(4):639-53. doi: 10.1016/j.eururo.2013.06.003. Epub 2013 Jun 12. PMID 23827737
- [Background] Ramsey EW, Elhilali M, Goldenberg SL, Nickel CJ, Norman R, Perreault JP, Piercy B, Trachtenberg J. Practice patterns of Canadian urologists in benign prostatic hyperplasia and prostate cancer. Canadian Prostate Health Council. J Urol. 2000 Feb;163(2):499-502. PMID 10647665
- [Background] Goldfischer ER, Cromie WJ, Karrison TG, Naszkiewicz L, Gerber GS. Randomized, prospective, double-blind study of the effects on pain perception of lidocaine jelly versus plain lubricant during outpatient rigid cystoscopy. J Urol. 1997 Jan;157(1):90-4. PMID 8976223
- [Background] Seklehner S, Remzi M, Fajkovic H, Saratlija-Novakovic Z, Skopek M, Resch I, Duvnjak M, Hruby S, Librenjak D, Hubner W, Breinl E, Riedl C, Engelhardt PF. Prospective multi-institutional study analyzing pain perception of flexible and rigid cystoscopy in men. Urology. 2015 Apr;85(4):737-41. doi: 10.1016/j.urology.2015.01.007. PMID 25817101
- [Background] Taghizadeh AK, El Madani A, Gard PR, Li CY, Thomas PJ, Denyer SP. When does it hurt? Pain during flexible cystoscopy in men. Urol Int. 2006;76(4):301-3. doi: 10.1159/000092051. PMID 16679829
- [Background] Song LJ, Lu HK, Wang JP, Xu YM. Cadaveric study of nerves supplying the membranous urethra. Neurourol Urodyn. 2010 Apr;29(4):592-5. doi: 10.1002/nau.20768. PMID 19760755
- [Background] Kozacioglu Z, Kiray A, Ergur I, Zeybek G, Degirmenci T, Gunlusoy B. Anatomy of the dorsal nerve of the penis, clinical implications. Urology. 2014 Jan;83(1):121-4. doi: 10.1016/j.urology.2013.07.075. Epub 2013 Nov 12. PMID 24238564
- [Background] Kirya C, Werthmann MW Jr. Neonatal circumcision and penile dorsal nerve block--a painless procedure. J Pediatr. 1978 Jun;92(6):998-1000. doi: 10.1016/s0022-3476(78)80386-2. PMID 660375
- [Derived] Qiu Y, Liu X, Wei W, Du G. Dorsal penile nerve block alleviates pain in men undergoing rigid cystoscopy: A single-center, randomized, double-blind, and placebo-controlled trial. BJUI Compass. 2021 Feb 5;2(4):260-266. doi: 10.1002/bco2.76. eCollection 2021 Jul. PMID 35475300
- [Derived] Qiu Y, Hu AM, Liu J, Du GZ. Dorsal penile nerve block for rigid cystoscopy in men: study protocol for a randomized controlled trial. Trials. 2016 Mar 18;17(1):147. doi: 10.1186/s13063-016-1281-9. PMID 26988368

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Started | 86 | 86 | 86
Completed | 86 | 86 | 86
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group | Total
Number analyzed (Participants) | 86 | 86 | 86 | 258
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (11.5) | 52.1 (13.0) | 53.5 (12.0) | 53.0 (12.2)
Sex/Gender, Customized [Number; unit: participants]
  Male | 86 | 86 | 86 | 258
Body weight [Mean (Standard Deviation); unit: Kg] | 66.8 (8.2) | 68.8 (9.6) | 66.4 (8.9) | 67.3 (8.9)
Height [Mean (Standard Deviation); unit: cm] | 167.3 (5.6) | 168.7 (5.5) | 167.8 (6.4) | 167.9 (5.8)
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] | 23.8 (2.4) | 24.2 (3.0) | 23.6 (2.7) | 23.8 (2.7)
Duration of cystoscopy [Mean (Standard Deviation); unit: min] | 3.5 (0.6) | 3.5 (0.5) | 3.4 (0.5) | 3.5 (0.6)
Cystoscopy history [Number; unit: participants]
  First-time cystoscopy | 60 | 58 | 61 | 179
  Repeat cystoscopy | 26 | 28 | 25 | 79

OUTCOME MEASURES:

1. Primary Outcome: Visual Analog Scale (VAS) for Pain
Description: A visual analog scale (VAS) ranging from 0 to 10 was used to assess the patients' pain during the procedure. 0 means no pain, 1 to 3 means mild pain, 4 to 7 means moderate pain, and 8 to 10 means severe pain. Patients were asked the VAS score to express the degree of pain at each time point.
Time Frame: at cystoscopic inspection of external sphincter
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
units on a scale | 6 [5 to 7] | 4 [3 to 6] | 4 [3 to 5]

2. Secondary Outcome: Visual Analog Scale (VAS) for Pain
Description: as for outcome 1
Time Frame: before gel administration
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Secondary Outcome: Visual Analog Scale (VAS) for Pain
Description: as for outcome 1
Time Frame: at cystoscopic inspection of penile and bulbar urethra
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
units on a scale | 1 [1 to 2] | 1 [1 to 2] | 1 [1 to 1]

4. Secondary Outcome: Visual Analog Scale (VAS) for Pain
Description: as for outcome 1
Time Frame: at cystoscopic inspection of prostate and bladder
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
units on a scale | 2 [0 to 2] | 0 [0 to 2] | 0 [0 to 1]

5. Secondary Outcome: Visual Analog Scale (VAS) for Pain
Description: as for outcome 1
Time Frame: after withdrawal of cystoscope
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Heart Rate Before Gel Administration
Time Frame: before gel administration
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
Beats per minute | 75.0 (9.7) | 75.9 (9.4) | 73.6 (10.2)

7. Secondary Outcome: Heart Rate at Cystoscopic Inspection of Penile and Bulbar Urthra
Time Frame: at cystoscopic inspection of penile and bulbar urethra
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
Beats per minute | 84.8 (11.7) | 83.8 (12.0) | 81.1 (10.4)

8. Secondary Outcome: Heart Rate at Cystoscopic Inspection of External Sphincter
Time Frame: at cystoscopic inspection of external sphincter
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
Beats per minute | 96.7 (14.1) | 90.2 (14.9) | 86.2 (10.9)

9. Secondary Outcome: Heart Rate After Withdrawal of Cystoscope
Time Frame: after withdrawal of cystoscope
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
Beats per minute | 76.7 (10.9) | 72.3 (10.0) | 71.6 (9.2)

10. Secondary Outcome: Mean Arterial Pressure Before Gel Administration
Time Frame: before gel administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
mmHg | 95.3 (10.2) | 96.6 (9.7) | 95.1 (9.9)

11. Secondary Outcome: Mean Arterial Pressure at Cystoscopic Inspection of Penile and Bulbar Urthra
Time Frame: at cystoscopic inspection of penile and bulbar urthra
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
mmHg | 100 (10.6) | 99.8 (10.1) | 98.2 (9.0)

12. Secondary Outcome: Mean Arterial Pressure at Cystoscopic Inspection of External Sphincter
Time Frame: at cystoscopic inspection of external sphincter
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
mmHg | 113.7 (11.7) | 105.8 (10.5) | 104.8 (9.2)

13. Secondary Outcome: Mean Arterial Pressure After Withdrawal of Cystoscope
Time Frame: after withdrawal of cystoscope
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
mmHg | 99.3 (9.8) | 95.7 (8.4) | 95.2 (8.6)

14. Secondary Outcome: Oxygen Saturation by Pulse Before Gel Administration
Time Frame: before gel administration
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
percentage | 99 [98 to 99] | 98 [97 to 99] | 99 [98 to 99]

15. Secondary Outcome: Oxygen Saturation by Pulse at Cystoscopic Inspection of Penile and Bulbar Urthra
Time Frame: at cystoscopic inspection of penile and bulbar urthra
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
percentage | 99 [98 to 99] | 98 [98 to 99] | 99 [98 to 99]

16. Secondary Outcome: Oxygen Saturation by Pulse at Cystoscopic Inspection of External Sphincter
Time Frame: at cystoscopic inspection of external sphincter
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
percentage | 99 [98 to 99] | 98 [97 to 99] | 99 [98 to 99]

17. Secondary Outcome: Oxygen Saturation by Pulse After Withdrawal of Cystoscope
Time Frame: after withdrawal of cystoscope
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
percentage | 99 [98 to 99] | 98 [98 to 99] | 99 [98 to 99]

18. Secondary Outcome: Breath Rate Before Gel Administration
Time Frame: before gel administration
Measure: Mean (Standard Deviation); unit: times per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
times per minute | 19.8 (1.1) | 19.6 (1.6) | 19.5 (1.3)

19. Secondary Outcome: Breath Rate at Cystoscopic Inspection of Penile and Bulbar Urthra
Time Frame: at cystoscopic inspection of penile and bulbar Urthra
Measure: Mean (Standard Deviation); unit: times per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
times per minute | 20.0 (1.2) | 19.8 (1.5) | 19.6 (1.3)

20. Secondary Outcome: Breath Rate at Cystoscopic Inspection of External Sphincter
Time Frame: at cystoscopic inspection of external sphincter
Measure: Mean (Standard Deviation); unit: times per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
times per minute | 20.1 (1.3) | 19.8 (1.7) | 19.8 (1.5)

21. Secondary Outcome: Breath Rate After Withdrawal of Cystoscope
Time Frame: after withdrawal of cystoscope
Measure: Mean (Standard Deviation); unit: times per minute
Arm/Group | Tetracaine Gel Group | Dorsal Penile Nerve Block Group | Combination Group
Number analyzed (Participants) | 86 | 86 | 86
times per minute | 19.7 (1.2) | 19.4 (1.5) | 19.4 (1.2)

ADVERSE EVENTS:
Time Frame: from beginning of dorsal penile nerve block to end of cystoscopy
Groups:
- Tetracaine Group: tetracaine gel plus DPNB with saline
- DPNB Group: DPNB with ropivacaine plus plain lubricant
- Combination Group: DPNB with ropivacaine plus tetracaine gel
Arm/Group | Tetracaine Group | DPNB Group | Combination Group
Serious Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/86
Other Adverse Events (participants affected / at risk) | 0/86 | 0/86 | 0/86

LIMITATIONS AND CAVEATS:
The VAS scale was the only main observe index, and patients could have different cognition of pain and this may affect the evaluation of pain.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No